CLINICAL TRIAL: NCT02872402
Title: Feasibility of a Lifestyle Intervention Early After Delivery on the Cardiometabolic Risk Profile of Women With Recent Gestational Diabetes
Brief Title: Feasibility of a Postpartum Lifestyle Intervention on the Cardiometabolic Risk Profile of GDM Women
Acronym: DEPART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Julie Robitaille, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEPART
Record Dates: First submitted 2016-08-04; First posted 2016-08-19 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Dietary Modification; Weight Loss; Physical Activity; Breastfeeding
Keywords: gestational diabetes; dietary modification; weight loss; physical activity; breastfeeding
MeSH Terms: conditions — Weight Loss; Motor Activity; Breast Feeding; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): At 2-mo postpartum, women will start the 1-yr lifestyle intervention that will consist of 7 face-to-face individual sessions of 1-hr (at 2, 3, 4, 5, 6, 9, 12 mo postpartum and a follow-up at 18 mo). Metabolic and anthropometric measurements will be assessed at 2,6,12 and 18 mo postpartum. In addition, 7 individual sessions of 30 min between face-to-face sessions will be carried out on the phone.
  Benefits of exclusive breastfeeding, healthy eating and physical activity will be portrayed at each visit .
  Interventions: Behavioral: Lifestyle intervention
- Active control lifestyle intervention (Active Comparator): Women in the control group will come to the testing unit at 2, 6, 12 and 18 mo postpartum for metabolic and anthropometric measurements and at 3, 4, 5, 9 mo for weight measurements only. They will receive standard lifestyle recommendations in the form of written information at each visit.
  Interventions: Behavioral: Active control lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Women who are still breastfeeding at the first postpartum visit will be encouraged to pursue. References to local breastfeeding supporting groups will be done, if needed. The intervention will be conducted in order to reach recommendations for food servings and nutrient needs. Particular attention will be paid to increase fruits, vegetables, fish and whole grains intake, and decrease added sugars and high fat meat/dairy products. Women will be strongly encouraged to be active at least 150 min/week. They will be provided with targeted strategies for exercising, types of exercises and tips for including physical activity into the daily routine as well as fun exercises for the whole family.
  Arms: Intervention group
Behavioral: Active control lifestyle intervention — Participants in the control group will receive standard lifestyle recommendations in the form of written information at each visit.
  Arms: Active control lifestyle intervention

SUMMARY:
The goal of the study is to investigate the effect of a lifestyle intervention program (adoption of exclusive breastfeeding, healthy diet and regular physical activity) on minimizing postpartum weight retention among women with recent GDM.

DETAILED DESCRIPTION:
Women with a history of gestational diabetes (GDM) are characterized by increased risk for subsequent type 2 diabetes (T2D) and cardiovascular disease (CVD). These women are also characterized by higher body mass index (BMI) and waist circumference compared to women without prior GDM. Failure to lose the weight gained during pregnancy can lead to increased BMI for subsequent pregnancies. As such, the childbearing-age period has been described as a potential period of weight gain and represents a critical window for the development of obesity, T2D and CVD. Therefore, strategies aiming at preventing postpartum weight retention (WR) and early cardiometabolic alterations in women with a history of GDM are of paramount importance. Principal investigator have shown that a low diet quality score was associated with greater adiposity and lower insulin sensitivity in women with prior GDM. Furthermore, less than 10% of women with prior GDM met the recommendations for breastfeeding, nutrition, and physical activity. Investigators have shown that attitude and perceived behavioral control were significant predictors of the intention to adopt healthy eating. For those who did engage in healthy behaviors, lower prevalence of cardiometabolic alterations was observed, providing supportive evidence that the adoption of healthy behaviors may be key to prevent the progression to an altered cardiometabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with GDM
* Fluent in French
* Had a singleton pregnancy
* At least 18 yrs old
* With a reported pre-pregnancy BMI ≥18.5 kg/m2

Exclusion Criteria:

* Women who had bariatric surgery
* Women who plan another pregnancy in the following year
* Women with a history of type 1 or type 2 diabetes
* Women with a multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Weight retention | 12 months postpartum

SECONDARY OUTCOMES:
Waist circumference | 12 months postpartum
Body composition | 12 months postpartum
Glucose | 12 months
Insuline | 12 months
Oral glucose tolerance test (75g) | 12 months
Glycated hemoglobin | 12 months
Lipid profile | 12 months
Resting blood pressure | 12 months
Breastfeeding duration | 12 months
  , time physically active
Healthy eating index | 12 months
Time physically active | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Robitaille, RD PhD, Principal Investigator — Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petitclerc I, Perron J, Dugas C, Mayer T, Raymond F, Di Marzo V, Veilleux A, Robitaille J. Association between gestational diabetes mellitus, maternal health and diet, and gut microbiota in mother-infant dyads. BMC Pregnancy Childbirth. 2025 Apr 24;25(1):486. doi: 10.1186/s12884-025-07584-2. PMID 40275186
- [Derived] Fradet A, Castonguay-Paradis S, Dugas C, Perron J, St-Arnaud G, Marc I, Doyen A, Flamand N, Dahhani F, Di Marzo V, Veilleux A, Robitaille J. The human milk endocannabinoidome and neonatal growth in gestational diabetes. Front Endocrinol (Lausanne). 2024 Jun 13;15:1415630. doi: 10.3389/fendo.2024.1415630. eCollection 2024. PMID 38938519
- [Derived] Dugas C, Laberee L, Perron J, St-Arnaud G, Richard V, Perreault V, Leblanc N, Marc I, Di Marzo V, Doyen A, Veilleux A, Robitaille J. Gestational Diabetes Mellitus, Human Milk Composition, and Infant Growth. Breastfeed Med. 2023 Jan;18(1):14-22. doi: 10.1089/bfm.2022.0085. Epub 2022 Nov 21. PMID 36409543